CLINICAL TRIAL: NCT06640816
Title: Effectiveness & Efficiency of Bupivacaine Regional Spinal Anesthesia in Non-ERACS and ERACS Caesarean Section Based on Height and BMI
Brief Title: Bupivacaine Effectivity and Efficiency for Regional Spinal Anesthesia in Non-ERACS and ERACS Caesarean Section
Status: Completed | Type: Observational
Sponsor: Universitas Jenderal Soedirman (Other)
Responsible Party: Principal Investigator, MM Rudi Prihatno, MD, Universitas Jenderal Soedirman
Other Study IDs: UJenderalSoedirman
Record Dates: First submitted 2024-09-25; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Patients with ASA Physical Status 1 - 2 Who Undergo Surgical Delivery (cesarean Section)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The most widely used regional anesthesia technique in Indonesia today is regional anesthesia with the subarachnoid (spinal) blockade method. In its development, this technique is not only used for surgery in the lower abdomen area, but also used as a management of acute pain. Especially for cases of pregnant patients undergoing cesarean section, in its development a method known as enhanced regional anesthesia for c-section (ERACS) emerged.

This technique is widely preferred by most patients. ERACS is considered very beneficial for patients, because this technique promises faster mobility after surgery with a longer duration of pain compared to conventional spinal regional anesthesia techniques.

The data collected from this study is secondary data derived from the medical records of patients in 2 private hospitals in Purbalingga Regency, which are taken and sorted systematically according to needs.

This study was conducted based on the situation and condition of health services in Indonesia which are highly dependent on state funding through the national health insurance system. The state funding emphasizes the effectiveness and efficiency of health services, including surgical and related procedures.

The question of this research :

1. Is Bupivacaine in ERACS patients better than Non-ERACS based on BMI and height?
2. Is Bupivacaine in ERACS patients more effective and efficient than Non-ERACS based on BMI and height?

DETAILED DESCRIPTION:
This study was conducted at 2 hospitals in Purbalingga Regency and is a routine procedure carried out by researchers since 2015 and collected gradually from January to December 2023. The purpose of this study was to see the effectiveness and efficiency of several standard procedures carried out by the author for several years on post-spinal anesthesia complications and the duration of mobilization. In general, the effectiveness and efficiency of an action will lead to costs. This study was divided into 4 groups, namely the dose group based on height and weight with the ERACS method (A1), the dose group based on height and weight non-ERACS (A2), the dose group not based on height and weight with the ERACS method (K1), and the dose group not based on height and weight non-ERACS (K2). The total sample used was 150 which was divided into 2, namely 100 cases based on height and weight and 50 cases not based on height and weight. The sampling technique used the purposive sampling method. The study was conducted during January - December 2023.

This study compared the effectiveness between groups as seen from postoperative hemodynamics (blood pressure and pulse), duration of pain relief, and the use of perioperative resuscitation drugs (ephedrine) based on the patient's height and weight. In patients in groups A1 and A2, the administration of 0.5% bupivacaine is when the height is > 150 cm, then the dose of bupivacaine is 10 mg and if the height is more than 160 cm, then the dose of bupivacaine is 15 mg. In groups K1 and K2, the administration of 0.5% bupivacaine is 20 mg. All statistical analyses were performed using IBM SPSS Statistics Software Version 20. The statistical tests used were the Wilcoxon Signed Ranks Test and the Kruskal Wallis Test adjusted to the needs and type of data. Data is considered significant if the p value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergo sectio caesaria
* ASA 1-2 phisically state

Exclusion Criteria:

- Patient refuses to participate

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant patients who come to the hospital and undergo delivery operations
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | Each patient's BMI is measured from the time they first come for antenatal care, until the patient goes home after giving birth (9 months)
  In Kg/ m2. BMI is an estimate of the ideal body weight for health. BMI does not measure body fat directly but is closely related to other measurements that measure body fat. BMI is calculated by dividing your weight in kilograms by the patients; height in square meters. BMI can be calculated using either metric or imperial (US) units. For imperial units, BMI is calculated by dividing your weight in pounds by your height in inches squared, then multiplying by 703.
Body weight | Each patient's body weight is measured from the time they first come for antenatal care, until the patient goes home after giving birth (9 months)
  Patient body weight in kilogram (Kg)
Body height | Measurements are taken once during pregnancy and also taken together with other measurements (BMI and bodyweight). Patients measured from the time they first come for antenatal care, until the patient goes home after giving birth (9 months)
  Patient height in meters

IPD SHARING:
Plan to Share IPD: Undecided
This study uses secondary data in Indonesian hospitals

REFERENCES:
- [Background] Huang Q, Wen G, Hai C, Zheng Z, Li Y, Huang Z, Huang B. A Height-Based Dosing Algorithm of Bupivacaine in Spinal Anesthesia for Decreasing Maternal Hypotension in Cesarean Section Without Prophylactic Fluid Preloading and Vasopressors: A Randomized-Controlled Non-Inferiority Trial. Front Med (Lausanne). 2022 Jun 10;9:858115. doi: 10.3389/fmed.2022.858115. eCollection 2022. PMID 35755061
- See also: Related Info — https://bmjopen.bmj.com/content/bmjopen/11/2/e040797/DC1/embed/inline-supplementary-material-1.pdf?download=true